CLINICAL TRIAL: NCT04233931
Title: Mhealth for Pre-exposure Prophylaxis Adherence by Young Adult MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Environment and Health Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1R43MH112221-01A1 (NIH)
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: pre-post test evaluation of the impact of a mobile app on PrEP treatment adherence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participant (Experimental): all participants in the study receive the mobile app.
  Interventions: Behavioral: PrEP medication adherence mobile app

INTERVENTIONS:
Behavioral: PrEP medication adherence mobile app — Participants use a PrEP medication adherence mobile app for six weeks.

SUMMARY:
The proposed project involves the development and testing of an mhealth intervention to increase adherence to PrEP treatment using texts providing tailored pill reminders, motivational messages, and health education messages. The intervention targets culturally-diverse young adult men who have sex with men (YMSM), who are at high risk for both HIV and non-adherence to PrEP medication. Supporting PrEP adherence would help reduce new HIV infections in this group.

DETAILED DESCRIPTION:
Specific Aims: Pre-exposure prophylaxis (PrEP) treatment greatly reduces HIV risk. When the PrEP pill (Truvada) is taken daily, it can reduce HIV risk up to 92%. NIH has designated reducing HIV/AIDS as a high-priority topic for research support using AIDS-designated funds. Among other groups, the CDC recommends PrEP for men who have sex with men (MSM) who are HIV-negative and in a relationship with an HIV+ partner, and MSM who have had anal sex without a condom or have been diagnosed with an STD in the past 6 months; about 1 in 4 MSM meet these criteria. Young people, age 13-29, accounted for 27% of new HIV cases in 2009. The highest concentration of new cases was among 20-29-year olds; 70% of these were MSM. Disparities are pronounced: 57% of new HIV cases reported in 2008-2010 were among African American MSM; 21% of cases were young Latino MSM. In PrEP trials to date, adherence has been generally low. Across these trials, younger age was the most consistent factor associated with lower PrEP adherence. Medication adherence can be difficult for young people. While young adults better comprehend benefits of prevention than teens, decision-making maturity is still developing through the 20s. It is not until the late 20s that two brain systems, one that spurs sensation-seeking and one that undergirds self-regulation and planning ahead, become integrated. Males may lag behind females in this regard. Furthermore, this developmental process can be hampered for those who have experienced the stress of victimization as have many MSM. PrEP adherence interventions for young adult MSM (YMSM) must take into account developmental factors that can affect decision-making. CDC strongly encourages PrEP prescribers to offer adherence support; foundational to that support is patient education. CDC also suggests adherence plans: 1) individually tailor dosing time 2) use pill reminders 3) use supports to address changes in routine and 4) consider disclosure issues, i.e. help patients identify social network members who can support adherence or ways to overcome adherence barriers due to lack of social disclosure. To date, no PrEP adherence intervention has been developed specifically for YMSM, despite increasing HIV rates in this group and their increased risk for non-adherence. High rates of texting by young adults, coupled with strong evidence base that text reminders can improve adherence, point to mobile health (mhealth) as an ideal way to support PrEP adherence among YMSM.

The goal of the proposed SBIR is to develop and test the feasibility and short-term effectiveness of an individually-tailored, developmentally- and culturally-sensitive mhealth PrEP adherence intervention for culturally-diverse YMSM. Its scientific premise rests on three large well-conducted adherence follow-up studies to PrEP efficacy trials, i.e. VOICE, FEM-PrEP, and iPrEx, which identified adherence facilitators/barriers being targeted in the proposed study, and on meta-analyses of a large and growing literature pointing to the effectiveness of mhealth for medication adherence across chronic conditions, including HIV. The intervention will be modeled on Dr Patricia Weitzman's (proposed PI) SBIR Phase 1 and 2 mhealth anti-retroviral therapy (ART) adherence intervention for HIV+ African Americans. That intervention employed a three-pronged approach of tailored pill reminders with age- and culturally-sensitive motivational and educational texts. Texts were designed to increase ART self-efficacy, and based on principles from social learning theory and positive psychology. Using a similar approach, formative research will be conducted to create motivational and educational texts that are culturally- and developmentally-sensitive for diverse YMSM. Moreover, formative research will allow us to identify and target unique PrEP adherence barriers and facilitators among culturally-diverse YMSM. Findings will be used to create and pilot a 6-week randomized mhealth PrEP adherence intervention addressing adherence barriers and facilitators identified in PrEP RCTs, and our formative research, as well as CDC PrEP adherence recommendations. Our long-term goal is to reduce HIV infection rates among culturally-diverse YMSM by supporting PrEP adherence.

Specific Aim 1: Develop a individually-tailored, culturally- and developmentally-sensitive mhealth intervention to promote adherence to PrEP among YMSM, ages 20-29. Aim 2: Implement 6-week pilot randomized controlled trial to evaluate short-term effectiveness (did it improve PrEP adherence, PrEP knowledge and PrEP treatment self- efficacy). CONSORT guidelines for the RCT will be followed in order to ensure scientific rigor. Primary Hypothesis: Young adult MSM who receive tailored daily pill reminder plus motivational/ educational texts for 6 weeks will show greater PrEP adherence compared to controls. Secondary Hypothesis: Young adult MSM who receive tailored daily pill reminder plus motivational/educational texts for 6 weeks will show greater PrEP knowledge and PrEP treatment self-efficacy compared to controls. Aim 3: Evaluate feasibility of the intervention, e.g. implementation fidelity (to what extent was intervention delivered as planned), program appeal (how well did participants like the intervention) and program reach (how well did it reach participants). CDC estimates PrEP is appropriate for the roughly 500,000 MSM in the US. Impact models show even modest adherence to PrEP could reduce new HIV infections among MSM by 29% over 20 years. An mhealth PrEP adherence tool targeting young adult MSM, a group experiencing increased HIV incidence, could not only support that reduction but-due to easy access and low cost-actually improve upon it.

ELIGIBILITY:
Inclusion criteria

* Male
* Age 20-29
* Currently taking PrEP
* Own smartphone

Exclusion criteria

* Current participation in PrEP or other HIV-related study
* Uncomfortable with potential privacy loss risks

Ages: 20 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self-identify as male
Enrollment: 54 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
PrEP medication adherence tool | 6 weeks
  A 3-item HIV medication adherence tool developed by Segeral was adapted for use with PrEP/Truvada to assess PrEP adherence

SECONDARY OUTCOMES:
PrEP treatment self-efficacy scale | 6 weeks
  The Adherence Self-Efficacy Scale developed by Johnson was adapted to assess participants' confidence to carry out PrEP treatment-related behaviors
PrEP knowledge Tool | 6 weeks
  PrEP knowledge Tool was developed by Weitzman and Kogelman to assess participants' knowledge of PrEP through questions about medication purpose, side effects, concomitant condom use, HIV testing
Intention to practice safe sex and adhere to 3-month follow-up HIV testing Tool | 6 weeks
  This tool was developed by Weitzman and Kogelman to assess participants' intention to practice safe sex and adhere to 3-month follow-up HIV testing recommendations for individuals on PrEP

CONTACTS AND LOCATIONS:
Overall Officials: patricia f weitzman, PhD, Principal Investigator — Environment and Health Group
Locations (1):
- Environment and Health Group, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We have no plan to make data available.